CLINICAL TRIAL: NCT03306381
Title: The Effect of Dietary Intervention on Symptoms in Relation to Genetical Characteristics, Epigenetics, Gut Microbiota, and Autoantibodies in IBS Patients
Brief Title: The Effect of Dietary Intervention on Symptoms, Epigenetics, and Gut Microbiota in IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IBS-2017
Record Dates: First submitted 2017-09-18; First posted 2017-10-11 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: IBS - Irritable Bowel Syndrome
Keywords: IBS; Epigenetics; Dietary intervention; Gut Microbiota; Inflammation; Genetics
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammation | interventions — Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention subject group (Experimental): n=130. Participants on low FODMAP-similar diet during 4-week study period.
  Interventions: Other: Dietary intervention
- Control group (No Intervention): n=20. Participants on traditional IBS diet during 4-week study period.

INTERVENTIONS:
Other: Dietary intervention — Elimination of certain products.
  Arms: Dietary intervention subject group

SUMMARY:
The aim of the present study is to research whether subjects with irritable bowel syndrome (IBS) display epigenetic/genetic changes or altered microbiota compared to a non-IBS control group. Further, we will investigate if these parameters as well as subjective IBS symptoms are affected by a 4-week long dietary intervention within the IBS patient group.

DETAILED DESCRIPTION:
The study will be performed on 140 subjects with verified IBS. Patients will be recruited from the clinic of Gastroenterology or Internal medicine as well as primary health care centers. At the start of the study patients will fill out protocols concerning Rom IV criteria (to validate that IBS criteria are filled) as well as IBS symptom rating scales. They will be examined by a physician/researcher who will complete protocols of clinical data. Blood and fecal samples will be collected. A control group of healthy, non-IBS individuals will go through the same procedure as described above.

Study participants with IBS will thereafter be randomized to receive an alternative diet resembling the FODMAP (Fermentable, Oligo-, Di-, Mono-saccharides And Polyols) diet (n=130), or to continue with their regular diet (control group; n=20). After 4 weeks of dietary intervention, there will be a follow-up where blood and fecal samples are once again collected. At this point in time, participants will also fill in IBS symptom rating scales again.

Samples from baseline and 4 weeks will be used for genetic/epigenetic (including genomic-wide association studies), gut microbiota and inflammatory parameter analyses.

Statistics

To study differences in the above-mentioned parameters between patients and controls as well as before and after dietary intervention, Mann-Whitney U-test and Wilcoxon test will be used, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Verified IBS according to Rom IV criteria.

Exclusion Criteria:

* Serious mental or somatic disease
* Abuse
* Inability to understand he Swedish language
* Already on a diet (e.g. vegan, FODMAP, gluten-free).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Genetic variation of enzymes regulating absorption of disaccharides | measured at baseline
  Genetic expression of disaccharide-degradating enzymes will be measured at baseline and related to the response of study participants to dietary intervention.

SECONDARY OUTCOMES:
Irritable bowel syndrome-subjective severity scores (IBS-SSS) ratings | 4 weeks
  Changes from baseline in subjective symptoms according to the IBS-SSS.
Visual analog scale for irritable bowel syndrome (VAS-IBS) ratings | 4 weeks
  Changes from baseline in subjective symptoms according to the VAS-IBS.
Gut microbiota composition | 4 weeks
  Changes from baseline in fecal microbiota analysed by 16rs
Cytokines | 4 weeks
  Changes from baseline in cytokine plasma concentrations will be assessed by ELISA.
microRNA expression | 4 weeks
  Changes from baseline in microRNA expression will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Bodil Ohlsson, MD, PhD, Principal Investigator — Region Skane
Locations (1):
- Deartment of INternal Medicine, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roth B, Ohlsson B. Overweight and vitamin D deficiency are common in patients with irritable bowel syndrome - a cross-sectional study. BMC Gastroenterol. 2024 Sep 3;24(1):296. doi: 10.1186/s12876-024-03373-x. PMID 39227769
- [Derived] Nilholm C, Manoharan L, Roth B, D'Amato M, Ohlsson B. A starch- and sucrose-reduced dietary intervention in irritable bowel syndrome patients produced a shift in gut microbiota composition along with changes in phylum, genus, and amplicon sequence variant abundances, without affecting the micro-RNA levels. United European Gastroenterol J. 2022 May;10(4):363-375. doi: 10.1002/ueg2.12227. Epub 2022 Apr 28. PMID 35484927